CLINICAL TRIAL: NCT04193189
Title: B-Enhancement of HBV Vaccination in Persons Living With HIV (BEe-HIVe): Evaluation of HEPLISAV-B
Acronym: BEe-HIVe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACTG A5379; 38569 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: HIV Infection; Hepatitis B
Keywords: vaccination; cytosine phosphoguanine adjuvant; seroprotection
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Heplisav-B; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A, 2-CpG: HEPLISAV-B (two injections) (Experimental): Participants were prescribed 0.5 mL of HEPLISAV-B (hepatitis B vaccine with a cytosine phosphoguanine adjuvant) by intramuscular (IM) injection at Weeks 0 and 4.
  Interventions: Biological: HEPLISAV-B
- Group A, 3-CpG: HEPLISAV-B (three injections) (Experimental): Participants were prescribed 0.5 mL of HEPLISAV-B (hepatitis B vaccine with a cytosine phosphoguanine adjuvant) by IM injection at Weeks 0, 4, and 24.
  Interventions: Biological: HEPLISAV-B
- Group A, 3-alum: ENGERIX-B (three injections) (Active Comparator): Participants were prescribed 1 mL of ENGERIX-B (conventional hepatitis B vaccine with an aluminum hydroxide adjuvant) by IM injection at Weeks 0, 4, and 24.
  Interventions: Biological: ENGERIX-B
- Group B: HEPLISAV-B (three injections) (Experimental): Participants were prescribed 0.5 mL of HEPLISAV-B (hepatitis B vaccine with a cytosine phosphoguanine adjuvant) by IM injection at Weeks 0, 4, and 24.
  Interventions: Biological: HEPLISAV-B

INTERVENTIONS:
Biological: HEPLISAV-B — Administered by IM injection
  Arms: Group A, 2-CpG: HEPLISAV-B (two injections); Group A, 3-CpG: HEPLISAV-B (three injections); Group B: HEPLISAV-B (three injections)
Biological: ENGERIX-B — Administered by IM injection
  Arms: Group A, 3-alum: ENGERIX-B (three injections)

SUMMARY:
The purpose of this study was to evaluate response to and safety of the HBV vaccine HEPLISAV-B in two study populations of people living with HIV: prior HBV vaccine recipients who are deemed non-responders and individuals who are naïve to HBV vaccination.

DETAILED DESCRIPTION:
This phase III/IV study evaluated the response to and safety of the HBV vaccine HEPLISAV-B in two study populations of people living with HIV: prior HBV vaccine recipients who are deemed non-responders (Group A) and individuals who are naïve to HBV vaccination (Group B). The analyses were conducted as separate evaluations of the two study populations for all primary and secondary objectives.

Group A (HBV vaccine non-responders)

The study was designed as an open-label three-arm study to evaluate whether:

1. HEPLISAV-B vaccination given as a two-dose series achieves non-inferior seroprotection response (SPR) compared to standard dose ENGERIX-B.
2. HEPLISAV-B vaccination given as a three-dose series achieves superior SPR compared to standard dose ENGERIX-B.

Participants were randomized in 1:1:1 ratio to the following study arms, stratified by sex at birth (male vs. female) and diabetes diagnosis status (yes vs. no):

2-CpG: Two doses of HEPLISAV-B at weeks 0 and 4.

3-CpG: Three doses of HEPLISAV-B at weeks 0, 4, and 24.

3-alum: Three doses of ENGERIX-B at weeks 0, 4, and 24.

The target sample size in Group A was 561 participants, 187 participants in each arm.

Group B (Naïve to HBV vaccination)

Group B study was a single arm evaluation of vaccine response and safety of three doses of HEPLISAV-B. The target sample size was 73 participants.

In both groups, participants were scheduled to attend several study visits through Week 72. All participants were to remain on their antiretroviral therapy (ART), not provided by the study, throughout the study. Visits included physical examinations and blood collection. For 7 days after each vaccination, participants were asked to record temperature and any reactions they experienced.

ELIGIBILITY:
Inclusion Criteria, Groups A and B

* HIV-1 infection
* On current HIV-1 antiretroviral therapy (ART)
* CD4+ T-cell count ≥100 cells/mm^3
* HIV-1 RNA <1000 copies/mL

Inclusion Criteria, Group A only

* Serum Hepatitis B antibody <10 mlU/mL, non-reactive (negative), or indeterminate
* Documentation of HBV vaccination >168 days prior to study entry

Inclusion Criterion, Group B only

* Serum Hepatitis B antibody non-reactive (negative) within 45 days prior to study entry

Exclusion Criteria, Groups A and B

* Infection or prior exposure to HBV
* Serum HBsAb level ≥10 mlU/mL or positive at screening or any other time prior to screening
* Presence of any active or acute AIDS-defining opportunistic infections
* Solid organ transplantation
* History of ascites, encephalopathy, or variceal hemorrhage
* Diagnosis of chronic kidney disease (CKD) stage G4
* Cancer diagnosis within 5 years
* Currently receiving chemotherapy
* Chronic use and/or receipt of systemically administered immunosuppressive
* Known allergy/sensitivity or any hypersensitivity to any HBV vaccine or yeast
* Active, serious infection other than HIV-1
* Receipt of any inactivated virus vaccine within 14 days
* Receipt of any of the following within 45 days prior to study entry:

  * Live virus vaccine
  * Granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF)
  * Any other investigational medicinal agent
* Receipt of immunoglobulin or blood products within 90 days prior to study entry
* Receipt of an injection of DNA plasmids or oligonucleotides within 60 days prior to study entry

Exclusion Criteria, Group A only

* Hepatitis B virus vaccination ≤168 days prior to study entry
* Receipt of HEPLISAV-B vaccine at any time prior to study entry

Exclusion Criterion, Group B only

* Known HBV vaccination prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Sherman, MD, PhD, Study Chair — Cincinnati CRS; Kristen Marks, MD, Study Chair — Weill Cornell Chelsea CRS
Locations (41):
- United States (28):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Whitman-Walker Health CRS, Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Weill Cornell Uptown CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Gaborone CRS, Gaborone, South-East District, Botswana
- Brazil (2):
  - Hospital Nossa Senhora da Conceicao CRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
- Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho, Rift Valley, Kenya
- Blantyre CRS, Blantyre, Malawi
- De La Salle Health Science Institute Angelo King Medical Research Center, Silang, Philippines
- South Africa (3):
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Perth Road, Westdene, Johannesburg, Gauteng
  - Durban International Clinical Research Site CRS, Durban, KwaZulu-Natal
  - Soweto ACTG CRS, Johannesburg, Soweto
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
- Joint Clinical Research Centre (JCRC)/Kampala Clinical Research Site, Kampala, Uganda
- Hanoi Medical University CRS, Đống Đa, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections network (ACTG) by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data.

REFERENCES:
- [Result] Marks KM, Kang M, Umbleja T, Avihingsanon A, Sugandhavesa P, Cox AL, Vigil K, Perazzo H, Price JC, Katsidzira L, Vernon C, Alston-Smith B, Sherman KE; ACTG 5379 Study Team. Immunogenicity and Safety of Hepatitis B Virus (HBV) Vaccine With a Toll-Like Receptor 9 Agonist Adjuvant in HBV Vaccine-Naive People With Human Immunodeficiency Virus. Clin Infect Dis. 2023 Aug 14;77(3):414-418. doi: 10.1093/cid/ciad201. PMID 37017075
- [Result] Marks KM, Kang M, Umbleja T, Cox A, Vigil KJ, Ta NT, Omoz-Oarhe A, Perazzo H, Kosgei J, Hatlen T, Price J, Katsidzira L, Supparatpinyo K, Knowles K, Alston-Smith BL, Rathod P, Sherman KE; ACTG 5379 (BEe-HIVe) Study Team. HepB-CpG vs HepB-Alum Vaccine in People With HIV and Prior Vaccine Nonresponse: The BEe-HIVe Randomized Clinical Trial. JAMA. 2025 Jan 28;333(4):295-306. doi: 10.1001/jama.2024.24490. PMID 39616603
- [Result] Kang M, Marks KM, Cox AL, Sherman KE. An efficient vaccine clinical trial: ACTG A5379 hepatitis B vaccine trial in persons with HIV. Vaccine. 2025 May 10;55:127028. doi: 10.1016/j.vaccine.2025.127028. Epub 2025 Mar 26. PMID 40147293
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/sites/default/files/daids-ae-grading-table-v2-nov2014.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from December 2020 to February 2023 at sites in USA and select countries in Africa, Asia and South America.
Groups:
- Group A: 2-CpG: Participants were prescribed 0.5 mL of HEPLISAV-B (hepatitis B vaccine with a cytosine phosphoguanine adjuvant) by intramuscular injection at Weeks 0 and 4.
- Group A: 3-CpG; Group B: Participants were prescribed 0.5 mL of HEPLISAV-B (hepatitis B vaccine with a cytosine phosphoguanine adjuvant) by intramuscular injection at Weeks 0, 4, and 24.
- Group A: 3-alum: Participants were prescribed 1 mL of ENGERIX-B (conventional 3-dose hepatitis B vaccine with an aluminum hydroxide adjuvant) by intramuscular injection at Weeks 0, 4, and 24.
Period: Overall Study
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Started | 187 | 189 | 187 | 75
Eligible Participants Who Initiated Study Vaccination (All analyses were limited to the participants who met the study eligibility criteria (subsequently referred to as "eligible participants") who initiated study vaccination series.) | 187 | 188 | 186 | 74
Completed (In Group B, one participant was found to have been ineligible after enrollment (reason not completed is shown as protocol violation).) | 176 | 179 | 176 | 74
Not Completed | 11 | 10 | 11 | 1
Not completed — Lost to Follow-up | 9 | 7 | 9 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants who initiated study vaccination series.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B | Total
Number analyzed (Participants) | 187 | 188 | 186 | 74 | 635
Age, Customized [Count of Participants; unit: Participants]
  18-26 years | 42 | 34 | 32 | 4 | 112
  27-39 years | 30 | 35 | 33 | 14 | 112
  40-49 years | 30 | 45 | 42 | 30 | 147
  50-59 years | 58 | 53 | 43 | 19 | 173
  ≥60 years | 27 | 21 | 36 | 7 | 91
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender identity by self report.
  Participants
    Cisgender | 184 | 181 | 180 | 72 | 617
    Transgender spectrum | 3 | 6 | 5 | 2 | 16
    Not reported | 0 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth.
  Participants
    Female | 67 | 68 | 67 | 40 | 242
    Male | 120 | 120 | 119 | 34 | 393
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 42 | 40 | 11 | 132
  Not Hispanic or Latino | 148 | 145 | 144 | 63 | 500
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 0 | 4
  Asian | 29 | 35 | 33 | 49 | 146
  Black or African American | 85 | 76 | 74 | 12 | 247
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  White | 62 | 62 | 72 | 11 | 207
  Other | 2 | 4 | 1 | 0 | 7
  Multiple | 2 | 1 | 2 | 0 | 5
  Unknown | 6 | 8 | 3 | 1 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 10 | 13 | 12 | 0 | 35
  United States | 103 | 102 | 107 | 20 | 332
  Malawi | 5 | 5 | 6 | 0 | 16
  Botswana | 10 | 9 | 10 | 0 | 29
  Brazil | 13 | 13 | 11 | 0 | 37
  South Africa | 14 | 12 | 11 | 6 | 43
  Uganda | 5 | 5 | 4 | 0 | 14
  Kenya | 8 | 8 | 5 | 0 | 21
  Thailand | 18 | 17 | 19 | 48 | 102
  Philippines | 1 | 4 | 1 | 0 | 6
CD4 cell count [Count of Participants; unit: Participants]
  <200 cells/mm^3 | 6 | 3 | 6 | 1 | 16
  200-<350 cells/mm^3 | 19 | 13 | 11 | 10 | 53
  350-<500 cells/mm^3 | 35 | 28 | 34 | 11 | 108
  ≥500 cells/mm^3 | 127 | 144 | 135 | 52 | 458
HIV-1 RNA [Count of Participants; unit: Participants]
  <40 copies/mL | 175 | 176 | 175 | 68 | 594
  ≥40 copies/mL | 12 | 12 | 11 | 5 | 40
  Indeterminate | 0 | 0 | 0 | 1 | 1
Diabetes status [Count of Participants; unit: Participants]
  Diabetes | 25 | 23 | 26 | 7 | 81
  No diabetes | 162 | 165 | 160 | 67 | 554
Anti-HBs [Count of Participants; unit: Participants] — Antibody titer against hepatitis B surface antigen. Population: Eligible participants who initiated study vaccination series, and had anti-HBs results available at entry.
  Participants
    number analyzed (Participants) | 185 | 188 | 186 | 74 | 633
    <10 mIU/mL | 182 | 185 | 182 | 74 | 623
    ≥10 mIU/mL | 3 | 3 | 4 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Primary Seroprotection Response
Description: Primary seroprotection response was defined as antibody titer against hepatitis B surface antigen (anti-HBs) ≥10 mIU/mL at 8 weeks after 2-dose vaccination series and at 4 weeks after 3-dose vaccination series. If the completion of the vaccine series was delayed (a delay of ≤4 weeks was allowed), the trial protocol specified obtaining an antibody result at 8 weeks for the 2-dose series or at 4 weeks for the 3-dose series after vaccine completion for use in the primary outcome analysis. The study was designed separately for the two study populations (Groups A and B), and the analysis was conducted separately, as prespecified in the study protocol and Statistical Analysis Plan (SAP). In Group A, two-sided 97.5% confidence intervals (CI) were specified for the SPR differences between study arms (presented in the Statistical Analyses sections below). In Group B, two-sided 95% Wilson CI around the single-arm estimate was specified (presented in the Data Table below).
Time Frame: Week 12 in Group A 2-CpG, Week 28 in Group A 3-CpG and 3-alum and in Group B
Population: Eligible participants who initiated study vaccination series and had anti-HBs data available at the specified time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 174 | 169 | 165 | 68
percentage of participants | 93.1 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CI around the estimate is provided in the Data Table. | 99.4 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CI around the estimate is provided in the Data Table. | 80.6 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CI around the estimate is provided in the Data Table. | 100 [94.7 to 100]
Statistical Analysis 1: Comparison: Group A: 2-CpG vs Group A: 3-alum; Primary objective of Group A; Test type: Non-Inferiority — Pre-specified non-inferiority margin (2-CpG minus 3-alum): -10%; Common proportion difference = 12.5, 97.5% CI 2-sided [4.1 to 20.9] — Common SPR proportion (expressed as percentage of participants) difference (2-CpG minus 3-alum) with two-sided 97.5% Newcombe confidence interval stratified by sex at birth and diabetes status; Mantel-Haenszel weights were used
Statistical Analysis 2: Comparison: Group A: 3-CpG vs Group A: 3-alum; Primary objective of Group A; Test type: Superiority; Common proportion difference = 18.4, 97.5% CI 2-sided [10.4 to 26.2] — Common SPR proportion (expressed as percentage of participants) difference (3-CpG minus 3-alum) with two-sided 97.5% Newcombe repeated confidence interval stratified by sex at birth and diabetes status; Mantel-Haenszel weights were used
Statistical Analysis 3: Comparison: Group A: 2-CpG vs Group A: 3-CpG; Secondary objective of Group A; Test type: Superiority; Common proportion difference = 6.0, 97.5% CI 2-sided [-0.2 to 11.8] — Common SPR proportion (expressed as percentage of participants) difference (3-CpG minus 2-CpG) with two-sided 97.5% Newcombe confidence interval stratified by sex at birth and diabetes status; Mantel-Haenszel weights were used

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: The protocol required reporting of (1) Grade ≥2 AEs, (2) AEs that led to a change in study treatment regardless of grade, (3) AEs meeting serious AE (SAE) definition or expedited AE (EAE) reporting requirement, (4) Grade ≥1 local and systemic injection reactions within 7 days of any study vaccine injection, (5) medically attended adverse events (MAAE) regardless of grade, and (6) potential immune-mediated AEs regardless of grade. Grading was per DAIDS AE Grading Table (Version 2.1): Grade 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening) and 5 (death). DAIDS EAE Manual (V1.0) was used. Wilson method was used for confidence intervals.
Time Frame: From study entry to study discontinuation (Week 72 or premature discontinuation)
Population: Eligible participants who initiated study vaccination series
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 187 | 188 | 186 | 74
percentage of participants | 73.3 [66.5 to 79.1] | 77.7 [71.2 to 83.0] | 73.7 [66.9 to 79.5] | 87.8 [78.5 to 93.5]

3. Secondary Outcome: Percentage of Participants With Seroprotection Response
Description: Seroprotection response (SPR) was defined as antibody titer against hepatitis B surface antigen (anti-HBs) ≥10 mIU/mL. Study visit weeks are according to protocol-specified visit windows; anti-HBs results outside visit windows were not included. These are snapshots at scheduled visits irrespective of delayed vaccinations, unlike the visits defined in Primary Outcome 1. The study was designed separately for the two study populations (Groups A and B), and the analysis was conducted separately, as prespecified in the study protocol and Statistical Analysis Plan (SAP). In Group A, two-sided 97.5% confidence intervals (CI) were specified for the SPR differences between study arms (presented in the Statistical Analyses sections below). In Group B, two-sided 95% Wilson CIs around the single-arm estimates were specified (presented in the Data Table below).
Time Frame: Weeks 4, 8, 12, 24, 28, 32 (Group A 3-CpG and 3-alum and Group B), 48 (Group A 3-CpG and 3-alum and Group B), 52 (Group A 2-CpG) and 72. The visit schedule differed between the study arms.
Population: Eligible participants who initiated study vaccination series, and had anti-HBs data available at the given time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 187 | 188 | 186 | 74
percentage of participants
  Week 4: SPR: number analyzed (Participants) | 177 | 177 | 174 | 73
  Week 4: SPR | 66.1 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 66.7 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 51.7 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 30.1 [20.8 to 41.4]
  Week 8: SPR: number analyzed (Participants) | 175 | 174 | 173 | 69
  Week 8: SPR | 89.1 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 90.8 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 64.2 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 87.0 [77.0 to 93.0]
  Week 12: SPR: number analyzed (Participants) | 172 | 169 | 167 | 72
  Week 12: SPR | 93.6 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 92.9 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 66.5 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 94.4 [86.6 to 97.8]
  Week 24: SPR: number analyzed (Participants) | 162 | 163 | 164 | 68
  Week 24: SPR | 95.1 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 95.0 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 61.6 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 98.5 [92.1 to 99.7]
  Week 28: SPR: number analyzed (Participants) | 163 | 162 | 160 | 68
  Week 28: SPR | 92.6 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 99.4 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 80.0 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 100 [94.7 to 100]
  Week 32: SPR: number analyzed (Participants) | 0 | 161 | 161 | 69
  Week 32: SPR |  | 98.8 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 74.5 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 100 [94.7 to 100]
  Week 48: SPR: number analyzed (Participants) | 0 | 168 | 160 | 70
  Week 48: SPR |  | 97.6 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 65.0 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 98.6 [92.3 to 99.7]
  Week 52: SPR: number analyzed (Participants) | 162 | 0 | 0 | 0
  Week 52: SPR | 89.5 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. |  |  |
  Week 72: SPR: number analyzed (Participants) | 159 | 161 | 153 | 71
  Week 72: SPR | 86.1 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 96.9 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 57.5 [NA to NA] — In Group A, CIs are provided for comparisons between study arms only (in the Statistical Analyses below), as specified in the study SAP. Group B is single-arm and CIs around the estimates are provided in the Data Table. | 97.2 [90.3 to 99.2]
Statistical Analysis 1: Comparison: Group A: 2-CpG vs Group A: 3-alum; Comparison of Group A 2-CpG and 3-alum at 4 weeks post last scheduled vaccination (Week 8 in 2-CpG, Week 28 in 3-alum); Test type: Superiority; Common proportion difference = 9.0, 97.5% CI 2-sided [0.1 to 18.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group A: 2-CpG vs Group A: 3-alum; Comparison of Group A 2-CpG and 3-alum at 8 weeks post last scheduled vaccination (Week 12 in 2-CpG, Week 32 in 3-alum); Test type: Superiority; Common proportion difference = 19.0, 97.5% CI 2-sided [10.0 to 27.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group A: 2-CpG vs Group A: 3-alum; Comparison of Group A 2-CpG and 3-alum at 24 weeks post last scheduled vaccination (Week 28 in 2-CpG, Week 48 in 3-alum); Test type: Superiority; Common proportion difference = 27.8, 97.5% CI 2-sided [17.7 to 37.2] — Common SP proportion (expressed as percentage of participants) difference (2-CpG minus 3-alum) with two-sided 97.5% Newcombe confidence interval stratified by sex at birth and diabetes status; Mantel-Haenszel weights were used
Statistical Analysis 4: Comparison: Group A: 2-CpG vs Group A: 3-alum; Comparison of Group A 2-CpG and 3-alum at 48 weeks post last scheduled vaccination (Week 52 in 2-CpG, Week 72 in 3-alum); Test type: Superiority; Common proportion difference = 32.3, 97.5% CI 2-sided [21.3 to 42.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group A: 3-CpG vs Group A: 3-alum; Comparison of Group A 3-CpG and 3-alum at 8 weeks post last scheduled vaccination (Week 32); Test type: Superiority; Common proportion difference = 23.8, 97.5% CI 2-sided [15.5 to 32.3] — Common SPR proportion (expressed as percentage of participants) difference (3-CpG minus 3-alum) with two-sided 97.5% Newcombe confidence interval stratified by sex at birth and diabetes status; Mantel-Haenszel weights were used
Statistical Analysis 6: Comparison: Group A: 3-CpG vs Group A: 3-alum; Comparison of Group A 3-CpG and 3-alum at 24 weeks post last scheduled vaccination (Week 48); Test type: Superiority; Common proportion difference = 32.3, 97.5% CI 2-sided [23.2 to 41.2] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 7: Comparison: Group A: 3-CpG vs Group A: 3-alum; Comparison of Group A 3-CpG and 3-alum at 48 weeks post last scheduled vaccination (Week 72); Test type: Superiority; Common proportion difference = 38.8, 97.5% CI 2-sided [28.9 to 48.1] — [estimate comment as in outcome 3, analysis 5]
Statistical Analysis 8: Comparison: Group A: 2-CpG vs Group A: 3-CpG; Comparison of Group A 3-CpG and 2-CpG at 4 weeks post last scheduled vaccination (Week 28 in 3-CpG, Week 8 in 2-CpG); Test type: Superiority; Common proportion difference = 10.0, 97.5% CI 2-sided [3.1 to 16.4] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 9: Comparison: Group A: 2-CpG vs Group A: 3-CpG; Comparison of Group A 3-CpG and 2-CpG at 8 weeks post last scheduled vaccination (Week 32 in 3-CpG, Week 12 in 2-CpG); Test type: Superiority; Common proportion difference = 4.8, 97.5% CI 2-sided [-0.8 to 10.5] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 10: Comparison: Group A: 2-CpG vs Group A: 3-CpG; Comparison of Group A 3-CpG and 2-CpG at 24 weeks post last scheduled vaccination (Week 48 in 3-CpG, Week 28 in 2-CpG); Test type: Superiority; Common proportion difference = 4.9, 97.5% CI 2-sided [-0.8 to 11.2] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 11: Comparison: Group A: 2-CpG vs Group A: 3-CpG; Comparison of Group A 3-CpG and 2-CpG at 48 weeks post last scheduled vaccination (Week 72 in 3-CpG, Week 52 in 2-CpG); Test type: Superiority; Common proportion difference = 7.2, 97.5% CI 2-sided [0.7 to 14.2] — [estimate comment as in outcome 1, analysis 3]

4. Secondary Outcome: Count of Participants by Anti-HBs Titer Categories
Description: Count of participants by antibody titer against hepatitis B surface antigen (anti-HBs), categorized using cutoffs at 5, 10, 100 and 1000 mIU/mL. The testing assay lower limit of quantitation was 5 mIU/mL and upper limit 1000 mIU/mL. Study visit weeks are according to protocol-specified visit windows; anti-HBs results outside visit windows were not included. Because high proportions of participants achieved anti-HBs above the assay upper limit of quantitation, the planned geometric mean analysis was not conducted. Instead, anti-HBs were summarized according to the categories shown in the Data Table below.
Time Frame: as for outcome 3
Population: Eligible participants who initiated study vaccination series, and had anti-HBs data available at the given time point
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 187 | 188 | 186 | 74
Participants
  Week 4: anti-HBs: number analyzed (Participants) | 177 | 177 | 174 | 73
  Week 4: anti-HBs: <5 mIU/mL | 47 | 52 | 80 | 46
  Week 4: anti-HBs: 5-9 mIU/mL | 13 | 7 | 4 | 5
  Week 4: anti-HBs: 10-99 mIU/mL | 34 | 46 | 36 | 10
  Week 4: anti-HBs: 100-1000 mIU/mL | 65 | 49 | 36 | 8
  Week 4: anti-HBs: >1000 mIU/mL | 18 | 23 | 18 | 4
  Week 8: anti-HBs: number analyzed (Participants) | 175 | 174 | 173 | 69
  Week 8: anti-HBs: <5 mIU/mL | 16 | 9 | 52 | 7
  Week 8: anti-HBs: 5-9 mIU/mL | 3 | 7 | 10 | 2
  Week 8: anti-HBs: 10-99 mIU/mL | 33 | 37 | 36 | 24
  Week 8: anti-HBs: 100-1000 mIU/mL | 72 | 68 | 46 | 28
  Week 8: anti-HBs: >1000 mIU/mL | 51 | 53 | 29 | 8
  Week 12: anti-HBs: number analyzed (Participants) | 172 | 169 | 167 | 72
  Week 12: anti-HBs: <5 mIU/mL | 8 | 6 | 47 | 4
  Week 12: anti-HBs: 5-9 mIU/mL | 3 | 6 | 9 | 0
  Week 12: anti-HBs: 10-99 mIU/mL | 39 | 38 | 42 | 19
  Week 12: anti-HBs: 100-1000 mIU/mL | 76 | 71 | 50 | 38
  Week 12: anti-HBs: >1000 mIU/mL | 46 | 48 | 19 | 11
  Week 24: anti-HBs: number analyzed (Participants) | 162 | 163 | 164 | 68
  Week 24: anti-HBs: <5 mIU/mL | 6 | 5 | 50 | 1
  Week 24: anti-HBs: 5-9 mIU/mL | 2 | 3 | 13 | 0
  Week 24: anti-HBs: 10-99 mIU/mL | 31 | 27 | 50 | 14
  Week 24: anti-HBs: 100-1000 mIU/mL | 85 | 79 | 42 | 34
  Week 24: anti-HBs: >1000 mIU/mL | 38 | 49 | 9 | 19
  Week 28: anti-HBs: number analyzed (Participants) | 163 | 162 | 160 | 68
  Week 28: anti-HBs: <5 mIU/mL | 6 | 1 | 25 | 0
  Week 28: anti-HBs: 5-9 mIU/mL | 6 | 0 | 7 | 0
  Week 28: anti-HBs: 10-99 mIU/mL | 29 | 6 | 28 | 2
  Week 28: anti-HBs: 100-1000 mIU/mL | 81 | 28 | 43 | 9
  Week 28: anti-HBs: >1000 mIU/mL | 41 | 127 | 57 | 57
  Week 32: anti-HBs: number analyzed (Participants) | 0 | 161 | 161 | 69
  Week 32: anti-HBs: <5 mIU/mL |  | 2 | 31 | 0
  Week 32: anti-HBs: 5-9 mIU/mL |  | 0 | 10 | 0
  Week 32: anti-HBs: 10-99 mIU/mL |  | 8 | 27 | 2
  Week 32: anti-HBs: 100-1000 mIU/mL |  | 39 | 47 | 11
  Week 32: anti-HBs: >1000 mIU/mL |  | 112 | 46 | 56
  Week 48: anti-HBs: number analyzed (Participants) | 0 | 168 | 160 | 70
  Week 48: anti-HBs: <5 mIU/mL |  | 3 | 45 | 0
  Week 48: anti-HBs: 5-9 mIU/mL |  | 1 | 11 | 1
  Week 48: anti-HBs: 10-99 mIU/mL |  | 15 | 32 | 5
  Week 48: anti-HBs: 100-1000 mIU/mL |  | 70 | 48 | 25
  Week 48: anti-HBs: >1000 mIU/mL |  | 79 | 24 | 39
  Week 52: anti-HBs: number analyzed (Participants) | 162 | 0 | 0 | 0
  Week 52: anti-HBs: <5 mIU/mL | 12 |  |  |
  Week 52: anti-HBs: 5-9 mIU/mL | 5 |  |  |
  Week 52: anti-HBs: 10-99 mIU/mL | 39 |  |  |
  Week 52: anti-HBs: 100-1000 mIU/mL | 84 |  |  |
  Week 52: anti-HBs: >1000 mIU/mL | 22 |  |  |
  Week 72: anti-HBs: number analyzed (Participants) | 159 | 161 | 153 | 71
  Week 72: anti-HBs: <5 mIU/mL | 16 | 5 | 53 | 1
  Week 72: anti-HBs: 5-9 mIU/mL | 6 | 0 | 12 | 1
  Week 72: anti-HBs: 10-99 mIU/mL | 45 | 25 | 32 | 10
  Week 72: anti-HBs: 100-1000 mIU/mL | 77 | 76 | 39 | 32
  Week 72: anti-HBs: >1000 mIU/mL | 15 | 55 | 17 | 27

5. Secondary Outcome: Percentage of Participants With Grade ≥2 AEs Post-vaccination Adverse Events
Description: The protocol required reporting of (1) Grade ≥2 AEs, (2) AEs that led to a change in study treatment regardless of grade, (3) AEs meeting serious AE (SAE) definition or expedited AE (EAE) reporting requirement, (4) Grade ≥1 local and systemic injection reactions within 7 days of any study vaccine injection, (5) medically attended adverse events (MAAE) regardless of grade, and (6) potential immune-mediated AEs regardless of grade. This outcome is limited to the Grade ≥2 AEs that occurred within 4 weeks after any study vaccination. Grading was per DAIDS AE Grading Table (Version 2.1): Grade 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening) and 5 (death). DAIDS EAE Manual (V1.0) was used. Wilson method was used for confidence intervals.
Time Frame: From study vaccination initiation to 4 weeks after last study vaccination (Week 8 in Group A 2-CpG, Week 28 in Group A 3-CpG and 3-alum and Group B)
Population: Eligible participants who initiated study vaccination series
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 187 | 188 | 186 | 74
percentage of participants | 33.7 [27.3 to 40.7] | 45.7 [38.8 to 52.9] | 43.5 [36.6 to 50.7] | 48.6 [37.6 to 59.8]

6. Other Pre Specified Outcome: Percentage of Participants With Primary Seroprotection Response by Sex
Description: Subgroup analysis of the primary seroprotection response outcome measure (as described in the Primary Outcome Measure 1 above) by sex. Descriptive summary of the SPR by subgroups; the study was not powered for testing the success of HEPLISAV-B vaccination within subgroups.
Time Frame: Week 12 in Group A 2-CpG, Week 28 in Group A 3-CpG and 3-alum and in Group B
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 174 | 169 | 165 | 68
percentage of participants
  Among females: number analyzed (Participants) | 64 | 65 | 58 | 38
  Among females | 98.4 | 98.5 | 89.7 | 100
  Among males: number analyzed (Participants) | 110 | 104 | 107 | 30
  Among males | 90.0 | 100 | 75.7 | 100

7. Other Pre Specified Outcome: Percentage of Participants With Primary Seroprotection Response by Race
Description: Subgroup analysis of the primary seroprotection response outcome measure (as described in the Primary Outcome Measure 1 above) by race. Descriptive summary of the SPR by subgroups; the study was not powered for testing the success of HEPLISAV-B vaccination within subgroups.
Time Frame: Week 12 in Group A 2-CpG, Week 28 in Group A 3-CpG and 3-alum and in Group B
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
Number analyzed (Participants) | 174 | 169 | 165 | 68
percentage of participants
  Among Asian race: number analyzed (Participants) | 28 | 35 | 30 | 48
  Among Asian race | 96.4 | 100 | 80.0 | 100
  Among Black race: number analyzed (Participants) | 81 | 72 | 65 | 11
  Among Black race | 97.5 | 100 | 92.3 | 100
  Among White race: number analyzed (Participants) | 54 | 51 | 65 | 8
  Among White race | 90.7 | 98.0 | 67.7 | 100
  Among Other or Unknown race: number analyzed (Participants) | 11 | 11 | 5 | 1
  Among Other or Unknown race | 63.6 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: From study entry to study discontinuation (Week 72 or premature discontinuation)
Description: Protocol required reporting of (1) Grade ≥2 AEs, (2) AEs that led to a change in study treatment regardless of grade, (3) AEs meeting SAE definition or EAE reporting requirement, (4) Grade ≥1 local and systemic injection reactions within 7 days of any study vaccine injection, (5) MAAEs regardless of grade, (6) potential immune-mediated AEs regardless of grade. DAIDS AE Grading Table (V2.1) and EAE Manual (V1.0) were used. Eligible participants who initiated study vaccination series are included.
Arm/Group | Group A: 2-CpG | Group A: 3-CpG | Group A: 3-alum | Group B
All-Cause Mortality (participants affected / at risk) | 1/187 | 1/188 | 0/186 | 0/74
Serious Adverse Events (participants affected / at risk) | 12/187 | 15/188 | 11/186 | 4/74
Other Adverse Events (participants affected / at risk) | 133/187 | 146/188 | 134/186 | 64/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: 2-CpG (N=187) | Group A: 3-CpG (N=188) | Group A: 3-alum (N=186) | Group B (N=74)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: 2-CpG (N=187) | Group A: 3-CpG (N=188) | Group A: 3-alum (N=186) | Group B (N=74)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Inner ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 1 | 1 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 4 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2 | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 3 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 3 | 4 | 0
Chills (General disorders) | 3 | 1 | 2 | 0
Chronic fatigue syndrome (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 27 | 33 | 33 | 19
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 2 | 1 | 0
Influenza like illness (General disorders) | 1 | 1 | 0 | 1
Injection site erythema (General disorders) | 9 | 15 | 16 | 6
Injection site induration (General disorders) | 0 | 0 | 0 | 1
Injection site joint pain (General disorders) | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 47 | 75 | 41 | 31
Injection site swelling (General disorders) | 14 | 14 | 15 | 6
Malaise (General disorders) | 22 | 34 | 26 | 19
Mass (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 3 | 2 | 6 | 1
Peripheral swelling (General disorders) | 1 | 1 | 3 | 0
Pyrexia (General disorders) | 9 | 11 | 9 | 8
Vaccination site joint pain (General disorders) | 0 | 0 | 0 | 1
Vaccination site pain (General disorders) | 1 | 0 | 0 | 4
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Allergy to chemicals (Immune system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 0 | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 14 | 12 | 14 | 16
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Cervicitis gonococcal (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 1 | 0
Dermatophytosis (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0
Endometritis (Infections and infestations) | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Fungal foot infection (Infections and infestations) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 3 | 0 | 1
Genital herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Groin infection (Infections and infestations) | 0 | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Latent syphilis (Infections and infestations) | 1 | 0 | 2 | 0
Latent tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Malaria (Infections and infestations) | 1 | 0 | 1 | 0
Monkeypox (Infections and infestations) | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 3 | 4 | 0
Neurosyphilis (Infections and infestations) | 0 | 0 | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 2 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 2 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Parasitic gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngeal chlamydia infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Proctitis chlamydial (Infections and infestations) | 0 | 1 | 1 | 1
Proctitis gonococcal (Infections and infestations) | 2 | 3 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Secondary syphilis (Infections and infestations) | 1 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sexually transmitted disease (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Strongyloidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
Syphilis genital (Infections and infestations) | 0 | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 1
Tooth infection (Infections and infestations) | 2 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 11 | 7 | 0
Urethritis chlamydial (Infections and infestations) | 0 | 0 | 1 | 0
Urethritis gonococcal (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Vaginitis gardnerella (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic bone injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Shoulder fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Traumatic pain (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 4 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 5 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 2 | 0
Blood creatinine increased (Investigations) | 7 | 3 | 5 | 1
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 6 | 7 | 10 | 1
Blood phosphorus decreased (Investigations) | 2 | 2 | 1 | 0
Blood pressure increased (Investigations) | 2 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 1 | 1 | 1 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 2 | 0
Carbon dioxide decreased (Investigations) | 2 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 6 | 6 | 5 | 0
Glomerular filtration rate decreased (Investigations) | 4 | 7 | 8 | 7
Glomerular filtration rate increased (Investigations) | 2 | 0 | 0 | 0
Haemoglobin (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 4 | 8 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Treponema test positive (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 4 | 3 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 4 | 4 | 5 | 8
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 7 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 10 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 33 | 25 | 18
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 2 | 2 | 2
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 30 | 38 | 32 | 17
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 2 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Post-traumatic headache (Nervous system disorders) | 1 | 0 | 0 | 0
Radicular pain (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Tardive dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 1 | 1
Bipolar II disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Genital odour (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Scrotal mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine spasm (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 4 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulval ulceration (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 9 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 2 | 6
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tonsillar exudate (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Brachioradial pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 5 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Abortion induced (Surgical and medical procedures) | 0 | 0 | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Female sterilisation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Nerve block (Surgical and medical procedures) | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 5 | 1 | 4 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Vasoconstriction (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (4):
  • Study Protocol and Informed Consent Form: V3.0 (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT04193189/Prot_ICF_000.pdf
  • Study Protocol: Clarification Memo V3.0 (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT04193189/Prot_001.pdf
  • Study Protocol: Letter of Amendment V2.0 (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04193189/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT04193189/SAP_003.pdf